CLINICAL TRIAL: NCT05277454
Title: A Multicenter, Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-653 in Treatment of Patients With Advanced Malignant Solid Tumors and Tenosynovial Giant Cell Tumor
Brief Title: Clinical Study of HMPL-653 in Treatment of Advanced Malignant Solid Tumors and TGCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-653-00CH1
Record Dates: First submitted 2022-02-06; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-01

CONDITIONS: Advanced Malignant Solid Tumors; TGCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-653 open-label treatment arm (Experimental): Dose-escalation Stage:
  Participants will be treated with escalating doses of HMPL-653 to determine the MTD and RP2D.
  Dose-expansion Stage:
  Participants will be enrolled in the expansion stage to better characterize the safety, tolerability, PK variability, and preliminary efficacy of HMPL-653 in TGCT and specific advanced solid tumors.
  Interventions: Drug: HMPL-653

INTERVENTIONS:
Drug: HMPL-653 — Dose-escalation Stage:
  Several dose levels will be evaluated for HMPL-653. The participants will receive oral HMPL-653 single-dose evaluation and oral HMPL-653 QD continuously treatment in a therapeutic cycle of 28 days until reaching the criteria for the end of treatment.
  Dose-expansion Stage:
  The participants will receive HMPL-653 treatment （RP2D）until reaching the criteria for the end of treatment.

SUMMARY:
To evaluate the safety and tolerability of HMPL-653 in patients with advanced solid tumors who have failure of standard of care or can not tolerate standard of care or those with TGCT, and to determine the maximum tolerated dose (MTD) and/or the recommended phase II clinical study dose (RP2D) of HMPL-653 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Aged 18 to 75 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy at least 12 weeks.
5. Adequate bone marrow, liver and kidney function.

Exclusion Criteria:

1. Toxicity associated with previous antitumor therapy not recovered to ≤CTCAE grade 1；
2. Previous treatment with anti-CSF1R therapy and have progressive disease;
3. Receiving approved systematic antitumor therapy or in the treatment period of other interventional clinical study within 4 weeks prior to the first dose.
4. Patients with central nervous system (CNS) malignant tumor or malignant solid tumor with known CNS metastasis;
5. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose-Limiting Toxicities(DLTs) | up to 33 days
  To evaluate the safety and tolerability of HMPL-653 for dose escalation period
Maximum tolerated dose (MTD) | up to 12 months
  The Maximum tolerated dose of HMPL-653
Recommended phase II dose (RP2D) | up to 12 months
  Recommended phase II dose of HMPL-653

SECONDARY OUTCOMES:
Pharmacokinetic-Cmax | up to 9 weeks
  Peak concentration of Pharmacokinetic
Pharmacokinetic-Tmax | up to 9 weeks
  Time to peak concentration of Pharmacokinetic
Pharmacokinetic-Ctrough | up to 9 weeks
  Trough concentration of Pharmacokinetic
Pharmacokinetic-t1/2 | up to 9 weeks
  Terminal elimination half-life of Pharmacokinetic
Pharmacokinetic-AUC0-t | up to 9 weeks
  Area under the plasma concentration-time curve of Pharmacokinetic
Pharmacokinetic-AUC0-∞ | From first dose up to C3D1, estimated up to 9 weeks
  Area under the plasma concentration-time curve of Pharmacokinetic
Pharmacokinetic-AUC0-τ | up to 9 weeks
  Area under the plasma concentration-time curve of Pharmacokinetic
Pharmacokinetic-CL/F | up to 9 weeks
  Apparent clearance of Pharmacokinetic
Pharmacokinetic-Vz/F | up to 9 weeks
  Apparent volume of distribution in the terminal phase of Pharmacokinetic
Pharmacokinetic-AR | up to 9 weeks
  AUC-based accumulation coefficient of Pharmacokinetic
Objective response rate (ORR) | 12 months
  The incidence of confirmed complete response or partial response.
Progression-free survival (PFS) | 12 months
  The time from the first dose of study treatment to PD or death for any reason, whichever comes first.
Disease control rate (DCR) | 12 months
  The proportion of patients with confirmed CR or PR or stable disease (SD) as the best response, and the duration of SD needs to be ≥6 weeks.
Time to response (TTR) | 12 months
  The time from the first dose of HMPL-653 to the first objective response.
Duration of response (DoR) | 12 months
  The time from the first appearance of confirmed CR or PR to PD or death for any reason (whichever comes first), in the patients with objective response.
Overall survival (OS) | 24 months
  The time from the first dose of study treatment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Prof, Principal Investigator — Jilin Provincial Cancer Hospital
Locations (5):
- China (5):
  - Jilin Provincial Cancer Hospital, Changchun
  - Harbin Medical University Cancer Hospital, Harbin
  - Linyi Cancer Hospital, Linyi
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No